CLINICAL TRIAL: NCT05748392
Title: A Post-market, Multicenter, Prospective, Single-arm Study Evaluating Safety and Performance of the Veraflo™ Cleanse Choice Complete™ Dressing
Brief Title: 3M Veraflo™ Cleanse Choice Complete™ (VFCCC) Clinical Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No longer required.
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-015054
Record Dates: First submitted 2023-02-14; First posted 2023-02-28 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: WOUNDS INJURIES
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Veraflo™ Cleanse Choice Complete™ Dressing Use with Assessments (Other): Subject will have Veraflo™ Cleanse Choice Complete™ dressing applied and used per instructions for use. 3D imaging and wound / peri-wound skin characteristics will be taken during the treatment.
  Interventions: Device: Wound and per-wound assessments While using Device

INTERVENTIONS:
Device: Wound and per-wound assessments While using Device — 3D imaging and wound and per-wound skin characteristics will be conducted initially, at dressing changes and at end of treatment/study.

SUMMARY:
The purpose of this external clinical study is to demonstrate the safety and performance of the Veraflo™ Cleanse Choice Complete™ Dressing Kit which will be used in conjunction with the V.A.C.® Ulta™ Therapy Unit, utilizing V.A.C. Veraflo™ Therapy instillation functions.

ELIGIBILITY:
Inclusion Criteria

* Subject is at least 22 years old at time of consent.
* Subject OR Legal Authorized Representative is able to provide informed consent.
* Subject has been confirmed to have a chronic, acute, traumatic, sub-acute, or dehisced wound, partial-thickness burn, ulcer (such as diabetic, pressure or venous insufficiency), flap or graft.

Exclusion Criteria:

* Subject is pregnant prior to application of the initial dressing*

  *Women who have had surgical sterilization by a medically accepted method (i.e. tubal ligation, hysterectomy, or oophorectomy) or are post-menopausal, defined as not having menstruation for > 12 months will not be required to undergo pregnancy testing.
* Subject has been diagnosed with a malignancy in the wound.
* Subject has untreated osteomyelitis.
* Subject has an untreated systemic infection.
* Subject has active cellulitis in the peri-wound area.
* Subject has a known allergy or hypersensitivity to study materials: dressing(s), and/or dressing components such as acrylic or silicone adhesives or polyurethane.
* Subject has, in the opinion of the investigator, a clinically significant condition that would impair the Subject's ability to comply with the study procedures.
* Subject has had radiation directly to the wound area.
* Subject has been diagnosed with a major vascular deficit limiting arterial inflow to the wound region, as determined by the Investigator's interpretation of the Subject's medical history.
* Subject has necrotic tissue with eschar present. NOTE: After debridement of necrotic tissue and complete removal of eschar, Veraflo™ Therapy may be used.
* Subject is participating in another interventional clinical study or was enrolled in a clinical trial within the last 30 days of Visit 1.
* Subject has non-enteric or unexplored fistula.
* Subject has a wound with any unexplored tunneling present.
* Subject has inadequate hemostasis at the wound site, as determined by the investigator.
* Subject has a wound with non-protected exposed vessels, anastomotic sites, organ, or nerves.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
ADE/SADE | Up to 14 days
  Subject incidence of Adverse Device Events (ADEs) and Serious ADEs (SADEs) during the use of the device.

SECONDARY OUTCOMES:
Total Wound Area (%) | Up to 14 days
  Percent change in total wound area (%) from baseline to end-of-study.
Non-viable Tissue (%) | Up to 14 days
  Change in the percentage of non-viable tissue from baseline to end-of-study.
Total Wound Volume (%) | Up to 14 days
  Change in the percentage of total wound volume (%) from baseline to end-of-study.

OTHER OUTCOMES:
Debridement | Up to 14 days
  Subject incidence of bedside debridement.
  * Subject incidence of operating room debridement.
  * Number of avoided debridement procedures in the operating room based on physician assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- 3M, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No